CLINICAL TRIAL: NCT06303739
Title: Induction Protocol for Psilocybin-Assisted Therapy in Treatment-Resistant Depression (TRD): A Pilot Study
Brief Title: Psilocybin-Assisted Therapy in Treatment-Resistant Depression
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-1421
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Refractory Depression; Treatment Resistant Depression
Keywords: psilocybin; psychedelic; refractory depression; psychedelic-assisted therapy; treatment-resistant depression; TRD; depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of two groups and will receive either one single treatment of psilocybin-assisted therapy with follow-up therapy and assessments or two treatments spaced two weeks apart with follow-up therapy and assessments.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study and limitations of study staffing, only those conducting assessments and ratings throughout the study will be masked to the treatments. All others, including participants, therapists, investigators, and study coordinator, will not be masked to the number of treatments a participant receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Psilocybin Treatment (Experimental): Participants will be administered one dose of a 25mg capsule of psilocybin. This will be administered one time.
  Interventions: Drug: psilocybin
- Two Psilocybin Treatments (Active Comparator): Participants will be administered one dose of a 25mg capsule of psilocybin. Two weeks later, the participant will be administered one more dose of a 25mg capsule of psilocybin.
  Interventions: Drug: psilocybin

INTERVENTIONS:
Drug: psilocybin — 25mg of psilocybin administered during treatment session, accompanied by preparation before, integration after, and assistive therapy during the session.

SUMMARY:
The goal of this clinical trial is to test how well psilocybin-assisted therapy works in treating people with depression. The main questions this study aims to answer are:

* Does psilocybin with assisted therapy help improve symptoms for people with depression?
* How long do the effects of this treatment last?

Participants will:

* Take part in a couple of screening and preparation visits.
* Be given psilocybin in one or two treatment sessions.
* Attend a series of follow-up sessions over the following year.
* Complete forms and surveys to test how their symptoms have changed and what they thought of their experience.

Researchers will also compare whether one treatment or two treatments help improve symptoms more for participants.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) ranks fourth in global disease burden and has significant morbidity, mortality, societal and financial costs. However, few adequate and effective treatments exist with 60% of MDD patients not responding sufficiently to an initial oral antidepressant treatment. These patients who experience treatment resistant depression (TRD), defined as an intolerance or lack of response to two antidepressants of different classes, have limited treatment options beyond the antidepressant treatments that often yield insufficient results or relapse. Psilocybin, a novel treatment, has been found to relieve symptoms of TRD, but there are limited studies on specific dosing and long term treatment follow-up. In this study, the investigators will look closer at the effectiveness of one treatment with psilocybin versus two treatments with psilocybin, as well as the long term effectiveness over the first 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Willingness to comply with all study procedures and availability for the study.
* Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-V) diagnosis of major depressive disorder.
* Currently experiencing a major depressive episode, lasting at least 3 months
* Failure to respond or inability to tolerate at least 2 guideline-concordant pharmacological treatments from different pharmacologic classes during the current major depressive episode
* Good health evidenced by medical history and routine lab tests
* No central nervous system (CNS) or neurocognitive impairment
* Ability to take oral medication and to follow to the psilocybin-assisted therapy protocol
* Identified support person to accompany patient home after dosing
* Use of effective contraception throughout the study by those with child-bearing potential
* Use of condoms or other effective contraceptive methods by males with reproductive potential
* Fully vaccinated and up to date on vaccination against COVID-19, as defined by Center for Disease Control guidelines
* Following Lifestyle Considerations throughout study (no nicotine containing products in clinical unit, refrain from operating heavy machinery for the duration of treatment day, no more than two servings 8 hours prior to treatment, no psychoactive drugs 72 hours before treatment, refrain from consuming foods that would interfere with drug absorption, minimize interaction with household immunocompromised contacts)

Exclusion Criteria:

* Family history (first- or second-degree relatives) or diagnosis of bipolar disorder with psychotic features, schizophrenia, schizoaffective disorder, hallucinogen-induced psychosis, anti-social personality disorder, or other psychotic disorder.
* Borderline personality disorder, defined by DSM-V criteria, that in the judgement of the Investigator is likely to complicate the assessment of clinical response to study treatments or limits the patient's ability to comply with study procedures.
* Alcohol or other substance use disorder (except tobacco/nicotine) that has been active within the 6 months prior to enrollment.
* Recent use (within past 4 weeks) of esketamine, ketamine or classic hallucinogens (psilocybin-containing mushrooms or LSD) or use of psychedelics within the past 6 months or more than 10 times in lifetime.
* Participants with active suicidal ideation or plan with a Columbia Suicide Severity Rating Scale (C-SSRS) score greater than or equal to 4.
* Current active self-injurious behavior, requiring medical attention or per investigator discretion.
* Diagnosis of Obsessive-compulsive disorder or post-traumatic stress disorder.
* Within 72 hours of psilocybin administration, use of nicotine, alcohol, or other controlled substances.
* Current delirium, dementia, amnestic disorder, or other cognitive disorders.
* Any current or past medical or neurological illness (including chronic pain syndromes and/or history of cerebrovascular event (excluding migraine)) that, in the opinion of the investigator, may confound the interpretation of study assessments
* Known allergic reactions to components of psilocybin.
* Medically instability at screening, including hepatic, renal, circulatory, cardiac (arrhythmia, uncontrolled hypertension, systolic BP > 140 mmHg or diastolic BP > 90 mmHg, abnormal QTc), pulmonary or CNS (seizure disorder or treatment with antiepileptic drugs) impairment.
* Current pregnancy or lactation.
* Febrile illness in last 3 weeks.
* Current use or use within 4 weeks of psilocybin administration of Monoamine oxidase inhibitors (MAOIs), alcohol dehydrogenase inhibitors and antipsychotics (concomitant medications will be allowed per investigator discretion).
* Current treatment with buproprion greater than 300mg/day.
* Current use of tramadol.
* Prior participation in psilocybin-assisted therapy trial and or regular use of hallucinogens
* Treatment with another investigational drug or other intervention during study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in HAM-D-17 Scores between Baseline and 2 Weeks after Treatment | Baseline, 2 weeks
  The change in Hamilton Depression Rating Scale 17 item (HAM-D-17) scores between baseline and 2 weeks after treatment
  The HAM-D-17 is a 17-item questionnaire used to measure severity of depression. The score ranges from 0 to 52. Higher scores indicate more severe depression.
Change in QIDS SR-16 Scores between Baseline and 2 Weeks after Treatment | Baseline, 2 weeks
  The change between depression scores as reported by Quick Inventory of Depressive Symptomatology Short Response-16 (QIDS SR-16) scores between baseline and 2 weeks after treatment
  The QIDS SR-16 is a 16-item questionnaire used to measure severity of depression. The scores range from 0 to 45. Higher scores indicate more severe depression.
Number of Participants Achieving Remission 2 Weeks after Treatment | up to 2 weeks
  Number of participants achieving remission (defined as a HAM-D-17 score less than 10) 2 weeks after treatment
Number of Participants Achieving Response 2 weeks after treatment | up to 2 weeks
  Number of participants achieving response (defined as a HAM-D-17 score that has decreased by greater than or equal to 50 percent compared to baseline) 2 weeks after treatment

SECONDARY OUTCOMES:
Number of Participants Achieving Remission at 6 Weeks | up to 6 weeks
  Number of participants achieving remission (defined as a HAM-D-17 score less than 10) 6 weeks after treatment
Number of Participants Achieving Response at 6 Weeks | up to 6 weeks
  Estimate the number of participants achieving response (defined as a HAM-D-17 score that has decreased by greater than or equal to 50 percent compared to baseline) at 6 weeks after treatment
Number of Participants Achieving Remission at 3 Months | up to 3 months
  Number of participants achieving remission (defined as a HAM-D-17 score less than 10) 3 months after treatment
Number of Participants Achieving Response at 3 Months | up to 3 months
  Estimate the number of participants achieving response (defined as a HAM-D-17 score that has decreased by greater than or equal to 50 percent compared to baseline) at 3 months after treatment
Number of Participants Achieving Remission at 6 Months | up to 6 months
  Number of participants achieving remission (defined as a HAM-D-17 score less than 10) 6 months after treatment
Number of Participants Achieving Response at 6 Months | up to 6 months
  Estimate the number of participants achieving response (defined as a HAM-D-17 score that has decreased by greater than or equal to 50 percent compared to baseline) at 6 months after treatment
Number of Participants Achieving Remission at 9 Months | up to 9 months
  Number of participants achieving remission (defined as a HAM-D-17 score less than 10) 9 months after treatment
Number of Participants Achieving Response at 9 Months | up to 9 months
  Estimate the number of participants achieving response (defined as a HAM-D-17 score that has decreased by greater than or equal to 50 percent compared to baseline) at 9 months after treatment
Number of Participants Achieving Remission at 12 Months | up to 12 months
  Number of participants achieving remission (defined as a HAM-D-17 score less than 10) 12 months after treatment
Number of Participants Achieving Response at 12 Months | up to 12 months
  Estimate the number of participants achieving response (defined as a HAM-D-17 score that has decreased by greater than or equal to 50 percent compared to baseline) at 12 months after treatment
Time to Relapse in Participants Who Showed Remission at 2 weeks | up to 1 year after treatment
  Of the number of participants achieving remission (defined as a HAM-D-17 score less than 10) 2 weeks after treatment, the amount of time until a relapse occurring thereafter occurs.
  Relapse is defined as a HAM-D-17 score greater than or equal to 17 and will be measured up to the study follow-up visit at 1 year.
Time to Relapse in Participants Who Showed Response at 2 Weeks | up to 1 year after treatment
  Of the number of participants achieving remission (defined as a HAM-D-17 score that has decreased by greater than or equal to 50 percent compared to baseline) 2 weeks after treatment, the amount of time until a relapse occurring thereafter occurs.
  Relapse is defined as a HAM-D-17 score greater than or equal to 17 and will be measured up to the study follow-up visit at 1 year.
Change in HAM-D-17 Scores between Baseline and 6 Weeks after Treatment | Baseline, 6 weeks
  The change in HAM-D-17 scores between baseline and 2 weeks after treatment
  The HAM-D-17 is a 17-item questionnaire used to measure severity of depression. The score ranges from 0 to 52. Higher scores indicate more severe depression.
Change in HAM-D-17 Scores between Baseline and 3 Months after Treatment | Baseline, 3 Months
  The change in HAM-D-17 scores between baseline and 2 weeks after treatment
  The HAM-D-17 is a 17-item questionnaire used to measure severity of depression. The score ranges from 0 to 52. Higher scores indicate more severe depression.
Change in HAM-D-17 Scores between Baseline and 6 Months after Treatment | Baseline, 6 Months
  The change in HAM-D-17 scores between baseline and 2 weeks after treatment
  The HAM-D-17 is a 17-item questionnaire used to measure severity of depression. The score ranges from 0 to 52. Higher scores indicate more severe depression.
Change in HAM-D-17 Scores between Baseline and 9 Months after Treatment | Baseline, 9 Months
  The change in HAM-D-17 scores between baseline and 2 weeks after treatment
  The HAM-D-17 is a 17-item questionnaire used to measure severity of depression. The score ranges from 0 to 52. Higher scores indicate more severe depression.
Change in HAM-D-17 Scores between Baseline and 12 Months after Treatment | Baseline, 12 months
  The change in HAM-D-17 scores between baseline and 2 weeks after treatment
  The HAM-D-17 is a 17-item questionnaire used to measure severity of depression. The score ranges from 0 to 52. Higher scores indicate more severe depression.
Change in QIDS SR-16 Scores between Baseline and 6 Weeks after Treatment | Baseline, 6 weeks
  The change between depression scores as reported by QIDS SR-16 scores between baseline and 2 weeks after treatment
  The QIDS SR-16 is a 16-item questionnaire used to measure severity of depression. The scores range from 0 to 45. Higher scores indicate more severe depression.
Change in QIDS SR-16 Scores between Baseline and 3 Months after Treatment | Baseline, 3 Months
  The change between depression scores as reported by QIDS SR-16 scores between baseline and 2 weeks after treatment
  The QIDS SR-16 is a 16-item questionnaire used to measure severity of depression. The scores range from 0 to 45. Higher scores indicate more severe depression.
Change in QIDS SR-16 Scores between Baseline and 6 Months after Treatment | Baseline, 6 Months
  The change between depression scores as reported by QIDS SR-16 scores between baseline and 2 weeks after treatment
  The QIDS SR-16 is a 16-item questionnaire used to measure severity of depression. The scores range from 0 to 45. Higher scores indicate more severe depression.
Change in QIDS SR-16 Scores between Baseline and 9 Months after Treatment | Baseline, 9 Months
  The change between depression scores as reported by QIDS SR-16 scores between baseline and 2 weeks after treatment
  The QIDS SR-16 is a 16-item questionnaire used to measure severity of depression. The scores range from 0 to 45. Higher scores indicate more severe depression.
Change in QIDS SR-16 Scores between Baseline and 12 Months after Treatment | Baseline, 12 Months
  The change between depression scores as reported by QIDS SR-16 scores between baseline and 2 weeks after treatment
  The QIDS SR-16 is a 16-item questionnaire used to measure severity of depression. The scores range from 0 to 45. Higher scores indicate more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Robert K McClure, MD, Principal Investigator — Director of Interventional Psychiatry
Locations (1):
- UNC Chapel Hill Medical Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be provided beginning 9 and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Demyttenaere K, Van Duppen Z. The Impact of (the Concept of) Treatment-Resistant Depression: An Opinion Review. Int J Neuropsychopharmacol. 2019 Feb 1;22(2):85-92. doi: 10.1093/ijnp/pyy052. PMID 29961822
- [Background] Dold M, Kasper S. Evidence-based pharmacotherapy of treatment-resistant unipolar depression. Int J Psychiatry Clin Pract. 2017 Mar;21(1):13-23. doi: 10.1080/13651501.2016.1248852. Epub 2016 Nov 16. PMID 27848269
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Keller MB, Shapiro RW, Lavori PW, Wolfe N. Recovery in major depressive disorder: analysis with the life table and regression models. Arch Gen Psychiatry. 1982 Aug;39(8):905-10. doi: 10.1001/archpsyc.1982.04290080025004. PMID 7103679
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Carhart-Harris R, Giribaldi B, Watts R, Baker-Jones M, Murphy-Beiner A, Murphy R, Martell J, Blemings A, Erritzoe D, Nutt DJ. Trial of Psilocybin versus Escitalopram for Depression. N Engl J Med. 2021 Apr 15;384(15):1402-1411. doi: 10.1056/NEJMoa2032994. PMID 33852780
- [Background] Carhart-Harris RL, Bolstridge M, Rucker J, Day CM, Erritzoe D, Kaelen M, Bloomfield M, Rickard JA, Forbes B, Feilding A, Taylor D, Pilling S, Curran VH, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: an open-label feasibility study. Lancet Psychiatry. 2016 Jul;3(7):619-27. doi: 10.1016/S2215-0366(16)30065-7. Epub 2016 May 17. PMID 27210031
- [Background] Carhart-Harris RL, Bolstridge M, Day CMJ, Rucker J, Watts R, Erritzoe DE, Kaelen M, Giribaldi B, Bloomfield M, Pilling S, Rickard JA, Forbes B, Feilding A, Taylor D, Curran HV, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: six-month follow-up. Psychopharmacology (Berl). 2018 Feb;235(2):399-408. doi: 10.1007/s00213-017-4771-x. Epub 2017 Nov 8. PMID 29119217
- [Background] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667
- [Background] Gukasyan N, Davis AK, Barrett FS, Cosimano MP, Sepeda ND, Johnson MW, Griffiths RR. Efficacy and safety of psilocybin-assisted treatment for major depressive disorder: Prospective 12-month follow-up. J Psychopharmacol. 2022 Feb;36(2):151-158. doi: 10.1177/02698811211073759. PMID 35166158
- [Background] Barrett FS, Johnson MW, Griffiths RR. Validation of the revised Mystical Experience Questionnaire in experimental sessions with psilocybin. J Psychopharmacol. 2015 Nov;29(11):1182-90. doi: 10.1177/0269881115609019. Epub 2015 Oct 6. PMID 26442957
- [Background] Maclean KA, Leoutsakos JM, Johnson MW, Griffiths RR. Factor Analysis of the Mystical Experience Questionnaire: A Study of Experiences Occasioned by the Hallucinogen Psilocybin. J Sci Study Relig. 2012 Dec;51(4):721-737. doi: 10.1111/j.1468-5906.2012.01685.x. PMID 23316089
- [Background] Murphy R, Kettner H, Zeifman R, Giribaldi B, Kartner L, Martell J, Read T, Murphy-Beiner A, Baker-Jones M, Nutt D, Erritzoe D, Watts R, Carhart-Harris R. Therapeutic Alliance and Rapport Modulate Responses to Psilocybin Assisted Therapy for Depression. Front Pharmacol. 2022 Mar 31;12:788155. doi: 10.3389/fphar.2021.788155. eCollection 2021. PMID 35431912
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996